CLINICAL TRIAL: NCT03839498
Title: Phase II Study of Axitinib (AG-013736) With Evaluation of the VEGF-pathway in Metastatic, Recurrent or Primary Unresectable Pheochromocytoma/Paraganglioma
Brief Title: Study of Axitinib (AG-013736) With Evaluation of the VEGF-pathway in Pheochromocytoma/Paraganglioma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Antonio Fojo, Professor of Medicine at the Columbia University Medical Center, Dept of Med Hematology & Onc, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR5314
Record Dates: First submitted 2019-01-31; First posted 2019-02-15 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Pheochromocytoma; Paraganglioma
Keywords: Axitinib
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Axitinib (AG-013736) (Experimental): Subjects with Recurrent or Primary Unresectable Pheochromocytoma/Paraganglioma will receive 16 weeks of therapy (Axitinib), and be seen in clinic every 4 weeks to monitor therapy.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — Axitinib (AG-013736) is an oral, potent and selective inhibitor of vascular endothelial growth factor (VEGF) receptors 1, 2, and 3.
  Starting dose level 1: 5 mg every morning; 5 mg every evening. Dose level 2: 7 mg every morning; 7 mg every evening. Dose level 3: 10 mg every morning; 10 mg every evening. Dose level -1: 3 mg every morning; 3 every evening. Dose level -2: 2 mg every morning; 2 mg every evening.
  Axitinib is supplied as 1 and 5-mg tablets and is administered orally twice a day with or without food, each morning and evening (i.e., every 12 hours). Axitinib will be given as self-administered.
  Other Names: AG-013736

SUMMARY:
Primary Objective:

To determine the response rate (RR) of metastatic or locally advanced pheochromocytoma/paraganglioma to axitinib administered daily.

Secondary Objectives:

* Determine the progression-free survival.
* In an exploratory manner examine the extent of activation of the VEGFR pathway in pheochromocytoma/paraganglioma using a semi-quantitative immunohistochemistry assay and examine the relationship with response to therapy.
* Perform pharmacogenomics analyses of drug metabolism and transport proteins through germline DNA examination.

DETAILED DESCRIPTION:
The long-term survival for malignant pheochromocytoma/paraganglioma (PHEO/PGL) may be limited because of its hormonal effects as well as its aggressive behavior and dissemination, particularly in some hereditary PHEO/PGL. Although several therapeutic modalities have been used to palliate malignant PHEO/PGL, a continued search for new agents to address the malignancy is needed to improve outcomes. One approach is to utilize drugs that target signaling pathways leading to decreased proliferation and survival of cancer cells. Some data in the literature suggests that in malignant PHEO/PGL, VEGF seems to play a role in the biology of the cancer and thus, its inhibition could reduce tumor growth. Sunitinib and imatinib has been used in a limited number of malignant pheochromocytomas with varying responses. Axitinib was designed to inhibit VEGFR that participates in tumor angiogenesis. In order to determine the activity of axitinib in tumor and hormonal responses in malignant PHEO/PGL, it will be used as a single agent in this study. The combination of cyclophosphamide; vincristine and dacarbazine have been shown to produce partial responses in malignant PHEO/PGL. The majority of the patients may have already received this combination or will receive this combination chemotherapy in the future. The goal is to develop multiple lines of effective treatments for this disease.

ELIGIBILITY:
Inclusion Criteria

Adults with a confirmed pathologic diagnosis of pheochromocytoma/paraganglioma by a CUMC/NYPH laboratory when such tissue is available to confirm.

In the event that outside tissue is not available:

An outside pathology report confirms the diagnosis of Pheo/PGL, AND the patient has nuclear medicine imaging studies that would only be positive in an adult patient with a diagnosis of Pheo/PGL (F-DOPA, Dotatate, F-Dopamine or MIBG)

* Imaging confirmation of metastatic disease
* Measurable disease at the time of enrollment as per RECIST 1.1.
* A life expectancy of at least 3 months and ECOG performance status ≤ 2
* Age ≥ 18 years
* Information available or pending regarding possible genetic alterations that can explain the patient's pheochromocytoma/paraganglioma (mutations in SDHB, SDHV or VHL genes)
* Last dose of chemotherapy or experimental therapy more than 4 weeks (6 weeks in the case of nitrosourea) prior to enrollment date; 2 weeks if the last therapy was received as part of a "phase 0" or "exploratory IND" trial. Last surgery more than 4 weeks prior to enrollment, to allow for wound healing. Core biopsies or FNA will not require any waiting period
* Last radiotherapy treatment ≥ 4 weeks prior to starting treatment with this protocol and there must be sites of measurable disease that did not receive radiation
* Prior therapeutic MIBG is allowed
* Organ and marrow function as defined below:
* Total bilirubin ≤ 1.5 x ULN (upper limit of normal), unless the patient meets the criteria for Gilbert's Syndrome. The upper limit value for bilirubin for subjects with Gilbert's Syndrome is less than 3 mg/dl.

  o Note: A diagnosis of Gilbert's disease will be made in the presence of (1) unconjugated hyperbilirubinemia noted on several occasions; (2) normal results from CBC count, reticulocyte count, and blood smear; (3) normal liver function test results; and (4) an absence of other disease processes that can explain the unconjugated hyperbilirubinemia.
* AST ≤ 2.5 x ULN, ALT ≤ 2.5 x ULN
* Amylase and lipase equal to, or less than, the institutional ULN.
* Creatinine clearance ≥ 40 ml/min (estimated or measured creatinine clearance) or serum creatinine ≤ 1.6 mg/dl

  o Random urine protein < 20 mg/dL. If ≥ 20 mg/dL then a 24-hour urine protein collection will be performed to accurately demonstrate that the 24-hour total is <1000 mg, the level acceptable for enrollment on study
* Absolute neutrophil count ≥ 500/mm3
* Platelet count ≥ 50,000/ mm3
* Ability to understand and sign an informed consent document.
* Ability and willingness to follow the guidelines of the clinical protocol.
* Because the effects of chemotherapy on the developing human fetus are potentially harmful, women of childbearing potential and men who participate in the study must agree to use adequate contraception (hormonal or barrier methods) before, during the study and for a period of 3 months after the last dose of chemotherapy.

Exclusion Criteria

* Patients with pheochromocytoma/paraganglioma tumors potentially curable by surgical excision alone as determined by the Principal Investigator in discussions with the surgical consultants
* Patients who have large abdominal masses impinging on bowel or pulmonary masses with encroached vessels and a potential to bleed will be considered on case by case basis after careful consultation with multiple disciplines such as radiologists and surgeons with main intent being patient safety.
* Unstable hypertension defined as a systolic blood pressure >150 mm Hg or diastolic pressure > 90 mmHg despite optimal medical management.
* Untreated brain metastases (or local treatment of brain metastases within the last 3 months) due to the poor prognosis of these patients and difficulty ascertaining the cause of neurologic adverse events.
* Pregnancy, due to the possible adverse effects on the developing fetus.
* Lactating women who are breast-feeding due to the possibility of transmitting axitinib to the child.
* The presence of a second malignancy, other than squamous cell carcinoma of the skin or in situ cervical cancer because it will complicate the primary objective of the study. Cancer survivors who have been free of disease for at least one year can be enrolled in this study.
* Patients with evidence of a bleeding diathesis
* Patients must not have received prior therapy with a TKI. Prior TKI usage in pheochromocytoma affects the same pathway as axitinib.
* Gastrointestinal abnormalities including:

  * Inability to take oral medications
  * Requirement for intravenous alimentation
  * Prior surgical procedure affecting absorption including total gastric resection
  * Treatment for active peptic ulcer disease in the past 6 months
  * Active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy.
  * Malabsorption syndrome
* Current use or anticipated need for treatment with drugs that are known potent CYP3A4 inhibitors (i.e., grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir, and delavirdine).
* Current use or anticipated need for treatment with drugs that are known CYP3A4 or CYP1A2 inducers (i.e., carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampin, and St. John's wort).
* Requirement of anticoagulant therapy with oral vitamin K antagonists. Low-dose anticoagulants for maintenance of patency of central venous access devices or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.
* Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis.
* Any of the following within 12 months prior to study drug administration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack and within 6 months before study drug administration for deep vein thrombosis or pulmonary embolism.
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Response Rate (RR) | Up to 16 weeks
  This study is designed to determine the percentage of patients whose cancer shrinks or disappears after treatment.

SECONDARY OUTCOMES:
Progression-free survival | Duration of time from start of treatment to time of progression or death, whichever occurs first; an average of up to 12 months
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Fojo, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No